CLINICAL TRIAL: NCT03689465
Title: A Comparison of PTCy-ATG and ATG Strategy in Haploidentical HSCT for Acute Graft-versus-host Disease Prophylaxis
Brief Title: PTCy-ATG vs ATG in Haploidentical HSCT for Acute Graft-versus-host Disease Prophylaxis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTCy-ATG-2018
Record Dates: First submitted 2018-08-13; First posted 2018-09-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-09

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; posttransplantation cyclophosphamide; antithymocyte globulin; viral infection; graft-versus-host disease
MeSH Terms: conditions — Virus Diseases; Graft vs Host Disease | interventions — Mycophenolic Acid; Cyclosporins; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTCy-ATG group (Active Comparator): PTCy-ATG group refers to treatment with PTCy-ATG protocol as GVHD prophylaxis at a total dose of 4.5mg/kg ATG, a dose of 50mg/kg/d cyclophosphamide (CTX), a dose of 2.5mg/kg/d Ciclosporin A （CsA）, and a dose of 1.0g/d Mycophenolate Mofetil(MMF).
  Interventions: Drug: ATG; Drug: CTX; Drug: Mycophenolate Mofetil; Drug: Ciclosporin A (CsA)
- ATG group (Active Comparator): ATG group refers to treatment with ATG protocol as GVHD prophylaxis at a total dose of 7.5mg/kg ATG, a dose of 2.5mg/kg/d Ciclosporin A （CsA）, a dose of 1.0g/d Mycophenolate Mofetil(MMF) and methotrexate (MTX, on days +1, +3 and +6).
  Interventions: Drug: ATG; Drug: Mycophenolate Mofetil; Drug: Ciclosporin A (CsA); Drug: methotrexate (MTX)

INTERVENTIONS:
Drug: ATG — In PTCy-ATG group, ATG will be intravenously infused via a central venous catheter from day -3 until day -1 at a total dose of 4.5mg/kg. In ATG group, ATG will be intravenously infused via a central venous catheter from day -5 until day -2 at a total dose of 7.5mg/kg.
Drug: CTX — In PTCy-ATG group, CTX will be intravenously infused via a central venous catheter on day +4 at a dose of 50mg/kg/d.
  Arms: PTCy-ATG group
Drug: Mycophenolate Mofetil — In PTCy-ATG group, Mycophenolate Mofetil will be taken orally from day +5 with the dosage of 0.5g twice a day. The dosage will be halved from day +30. In ATG group, Mycophenolate Mofetil will be taken orally from day -9 with the dosage of 0.5g twice a day. The dosage will be halved from day +30.
Drug: Ciclosporin A (CsA) — In PTCy-ATG group, Ciclosporin A (CsA) will be intravenously infused from day +5 at a dose of 2.5mg/kg/d. In ATG group, Ciclosporin A (CsA) will be intravenously infused from day -9 at a dose of 2.5mg/kg/d.
Drug: methotrexate (MTX) — In ATG group, methotrexate (MTX) will be intravenously on days +1, +3 and +6.
  Arms: ATG group

SUMMARY:
The granulocyte colony-stimulating factor (G-CSF)+antithymocyte globulin (ATG)-based protocols and posttransplantation cyclophosphamide (PTCy) protocols have been widely used for graft-versus-host disease (GVHD) prophylaxis in haploidentical related donor transplantation (haplo-HSCT). Nevertheless, severe acute GVHD remains an obstacle for haplo-HSCT. This study is aim to evaluate the efficacy of a modified protocol that includes PTCY and ATG in recipients of haplo-HSCT.

DETAILED DESCRIPTION:
Haploidentical related donor transplantation is now considered an important alternative to allogeneic hematopoietic stem cell transplantation (allo-HSCT). Currently, the strategies for graft-versus-host disease (GVHD) prophylaxis mainly include ex vivo and in vivo T-cell depletion (TCD) in haploidentical HSCT (haplo-HSCT). In vivo TCD modalities have become mainstream including granulocyte colony-stimulating factor (G-CSF)+antithymocyte globulin (ATG)-based protocols and posttransplantation cyclophosphamide (PTCy) protocols. The ATG strategy has been widely used. Nevertheless, severe acute GVHD remains an obstacle for haplo-HSCT. In addition, infections, especially viral infections, remain an important drawback of this strategy. This study is aim to evaluate the efficacy of a modified protocol that includes PTCY and ATG in recipients of haplo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 18-65 years
* Haploidentical hematopoietic stem cell transplant recipient
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
CMV DNAemia | 1 year posttransplantation
  CMV DNAemia was defined as positive CMV-DNA in the blood when the copies exceeded 500 copies/ml.

SECONDARY OUTCOMES:
aGVHD | 100 days 1 year posttransplantation
  aGVHD (acute GVHD) was defined according to the 1994 Consensus Conference on Acute GVHD Grading and graded from I to IV.
cGVHD | 2 year posttransplantation
  Chronic GVHD (cGVHD) was graded as limited or extensive.
EBV DNAemia | 1 year posttransplantation
  EBV DNAemia was defined as positive EBV-DNA in the blood when the copies exceeded 500 copies/ml.
Leukemia relapse | 2 year posttransplantation
  primary disease relapse
OS | 2 year posttransplantation
  overall survival
DFS | 2 year posttransplantation
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (7):
- China (7):
  - Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Peking University People's Hospital, Beijing

REFERENCES:
- [Background] Wang Y, Fu HX, Liu DH, Xu LP, Zhang XH, Chang YJ, Chen YH, Wang FR, Sun YQ, Tang FF, Liu KY, Huang XJ. Influence of two different doses of antithymocyte globulin in patients with standard-risk disease following haploidentical transplantation: a randomized trial. Bone Marrow Transplant. 2014 Mar;49(3):426-33. doi: 10.1038/bmt.2013.191. Epub 2013 Dec 2. PMID 24292519
- [Background] Chang YJ, Huang XJ. Haploidentical SCT: the mechanisms underlying the crossing of HLA barriers. Bone Marrow Transplant. 2014 Jul;49(7):873-9. doi: 10.1038/bmt.2014.19. Epub 2014 Feb 24. PMID 24566712
- [Background] Baron F, Mohty M, Blaise D, Socie G, Labopin M, Esteve J, Ciceri F, Giebel S, Gorin NC, Savani BN, Schmid C, Nagler A. Anti-thymocyte globulin as graft-versus-host disease prevention in the setting of allogeneic peripheral blood stem cell transplantation: a review from the Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation. Haematologica. 2017 Feb;102(2):224-234. doi: 10.3324/haematol.2016.148510. Epub 2016 Dec 7. PMID 27927772